CLINICAL TRIAL: NCT00826904
Title: Regulation Of Maternal Fuel Supply And Neonatal Adiposity
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-0535; R56DK078645 (NIH)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Fetal Macrosomia; Gestational Diabetes
Keywords: Fetal programming; Fetal macrosomia; Fetal health; Gestational diabetes; Maternal health; Maternal obesity
MeSH Terms: conditions — Fetal Macrosomia; Diabetes, Gestational; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lean: Healthy, pregnant women with BMI of 20 - 26 kg/m2
- Obese: Healthy, obese pregnant women with BMI 30 - 38 kg/m2

SUMMARY:
The purpose of this study is to determine whether unrecognized maternal hyperglycemia and postprandial lipemia early or late in gestation predicts excess neonatal adiposity.

DETAILED DESCRIPTION:
Mounting epidemiologic evidence suggests that maternal obesity and Gestational Diabetes Mellitus (GDM) independently influence size at birth and disease susceptibility later in life. A major gap in the understanding of fetal programming is the knowledge of whether and how exposure to excess maternal fuels in the absence of frank hyperglycemia impacts fetal fat accretion. The investigators hypothesis is that neonatal adiposity results from unrecognized maternal hyperglycemia and excess lipid availability in gestation, in part caused by excessive lipolysis in the white adipose tissue of obese women, some of whom will be subsequently diagnosed as having GDM. In Aim 1 the investigators will test the hypothesis that in obese women, some of whom will later be diagnosed with GDM, increased lipolysis and unrecognized hyperglycemia and hypertriglyceridemia occur earlier in gestation than in lean women, resulting in increased plasma non-esterified fatty acids (NEFA), glycerol, triglycerides (TGs), and glucose available for fetal metabolism. In Aim 2 the investigators will test the hypothesis that fetal adiposity by ultrasound and neonatal adiposity by Dual-energy X-ray Absorptiometry (DXA) are strongly correlated with excess lipid and glucose availability in obese mothers early in gestation, regardless of GDM status, and that fasting biomarkers of neonatal insulin sensitivity will correlate with neonatal adiposity. In Aim 3 the investigators will test the hypothesis that the in-vitro suppression of lipolysis in white adipose tissue correlates with excess NEFA and TG availability in-vivo and is predictive of neonatal adiposity. The elucidation of specific derangements in both glucose and lipid metabolism and their timing in gestation in mothers who deliver infants with excess adiposity could challenge our current screening methods and entirely redirect our treatment to target the responsible maternal fuels. On a public health level, this research is instrumental to the investigators understanding of how an intrauterine environment may deliver excess glucose and/or lipids to the fetus and contribute to the genesis of the pediatric obesity epidemic. Such information may result in new treatment strategies in pregnant women to normalize fetal growth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 yr
* Pregnant (12-14 weeks gestation)
* Lean (BMI 20-26 kg/m2)
* Obese (BMI 30-38 kg/m2)

Exclusion Criteria:

* Age < 18 or > 35 yr
* Pre-existing diabetes
* Chronic medical conditions:

  1. hypertension,
  2. hepatitis,
  3. Human immunodeficiency Virus (HIV),
  4. Thrombophilias,
  5. History of:

     1. thromboembolism,
     2. renal disease,
     3. neurologic diseases,
     4. rheumatologic disorders,
     5. gastrointestinal disease,
     6. cardiac dysfunction, or
     7. pulmonary disease
* Obstetric conditions:

  1. history of stillbirth,
  2. severe growth restriction,
  3. severe preeclampsia, or
  4. placental abruption
* Medications known to affect lipid or glucose metabolism:

  1. Metformin,
  2. glucocorticoids,
  3. beta agonists or blockers, or
  4. antihypertensives
* Use of recreational drugs, alcohol or tobacco.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lean (BMI 20-26 kg/m2)and Obese (BMI 30-38 kg/m2) pregnant women (age 18-35 yr) without chronic medical conditions or obstetric complications will be enrolled at 12-14 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2007-10; Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Change in neonatal adiposity by maternal Triglycerides, Glucose | 14-16, 26-28 weeks gestation
  Prediction of neonatal adiposity by maternal Triglycerides and Glucose
Change in maternal postprandial lipemia | 26-28 weeks gestation

SECONDARY OUTCOMES:
Change in maternal postprandial lipemia | 14-16, 26-28 weeks gestation
Change in maternal postprandial glycemia | 14-16, 26-28 weeks gestation
Prediction of neonatal adiposity by placental and maternal adipose tissue lipoprotein lipase (LPL) activity | 26-28 weeks gestation
  adipose tissue biopsy/Neonatal adiposity by Dual x-ray Absorptiometry (DXA)
Correlation of neonatal adiposity and fetal growth | 28-30 weeks gestation
  Neonatal adiposity by Dual-energy X-ray Absorptiometry (DXA)
Correlation of neonatal adiposity and fetal growth | 36-37 weeks gestation
  Neonatal adiposity by Dual-energy X-ray Absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Barbour, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbour LA, Farabi SS, Friedman JE, Hirsch NM, Reece MS, Van Pelt RE, Hernandez TL. Postprandial Triglycerides Predict Newborn Fat More Strongly than Glucose in Women with Obesity in Early Pregnancy. Obesity (Silver Spring). 2018 Aug;26(8):1347-1356. doi: 10.1002/oby.22246. Epub 2018 Jun 22. PMID 29931812